CLINICAL TRIAL: NCT06680843
Title: Characterization of Human Immune Signatures to Zoonotic Virus Exposure in Cambodia
Acronym: Camzoo
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 002014
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Immunity, Humoral

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Whole blood collection — 30 mL at Day 0 with optional visits for up to 2 additional whole blood collections at least 30 days apart

SUMMARY:
This is a biospecimen procurement protocol to characterize the immune response to zoonotic virus exposure in healthy adult humans aged 18 to 65 years with high-risk exposure to animals or their excreta (e.g., guano farming and wet markets), or living within 5 km of animal habitats (e.g., bat caves and bat roosts) in Cambodia.

DETAILED DESCRIPTION:
This is a biospecimen procurement protocol to characterize immune signatures to zoonotic virus exposure in healthy adult humans aged 18 to 65 years who handle suspected infected animals or their excreta, or living within 5 km of animal reservoirs, in Cambodia.

The primary study objective is to characterize immunity to zoonotic viruses, specifically H5N1. To meet this objective, when possible, individuals with the highest likelihood of prior exposure to the viruses of interest (Nipahvirus, bCoVs, H5N1) will be screened for study inclusion. These high-exposure risk behaviors include direct handling of known or suspected infected animals or their excreta. If insufficient individuals meeting these criteria are found, then sampling will include individuals with lower risk exposures, including living or working in areas proximal to (within 5 km of) animal habitats.

All human subjects research activities will be conducted by study personnel within the International Center of Excellence in Research Cambodia, Cambodian CCDC, and the Forestry Administration of the Royal Government of Cambodia. NIH investigators are involved in study design, implementation, analysis of coded samples and data, and writing and dissemination of reports of study results. Although they may support Cambodian investigators in monitoring/oversight capacities, NIH investigators will not be engaged in human subjects research.

ELIGIBILITY:
Inclusion Criteria:

1. Capacity to provide informed consent.
2. Adult aged 18-65 years.
3. Have interaction with suspected infected animals within the last 2 years, including (but not limited to) the following risk factors:

   1. Hunting, slaughtering, or consuming suspected infected animals;
   2. Fruit collection, date palm sap harvesting, or tree pruning within agricultural plantations containing bat roosts;
   3. Bat guano farming;
   4. Ancillary work in live animal markets or wild animal habitats identified as likely containing infected animals (e.g., provision of cleaning, transportation, or tourism services);
   5. Living within 5 km of identified animal markets or wild animal habitats identified as likely containing infected animals.
4. Willing to allow biological samples and data to be stored for future research.

Exclusion Criteria:

1. Pregnancy (based on self-reporting).
2. Any underlying, chronic, or current medical condition that, in the opinion of the investigator, would interfere with participation in the study (e.g., inability or great difficulty in drawing blood, known anemia).
3. Self-reported symptoms suggestive of acute infection (acute myalgias, arthralgias, headache, retro-orbital pain, dyspnea, rash) within 7 days prior to enrollment.
4. Signs suggestive of acute infection (fever, defined as internal temperature >38°C; hypoxemia, defined as peripheral oxygen saturation of <90%; hypotension, defined as systolic blood pressure <90 mm Hg or diastolic blood pressure <50 mm Hg) present at screening.
5. Self-reported diagnosis of immune deficiency, including HIV infection, chronic corticosteroid use (≥10 mg prednisone dose or its equivalent for a continuous period of ≥30 days within the last 1 year), ongoing or prior (within the last 10 years) receipt of chemotherapy or immunotherapy, or current hematological malignancy.
6. Receipt of blood products, including immunoglobulin products, within 120 days of study enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults aged 18 to 65 years who handle suspected infected animals or their excreta, or living within 5 km of animal reservoirs, in Cambodia (n=160 to 320).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Antibody binding activity in plasma samples against known immunodominant zoonotic viral proteins | Day 0 and 2 optional visits at least 30 days apart between Day 180-720
  Measured by binding antibody titer greater than cutoffs established from healthy U.S. donors (3 standard deviations above mean signal intensity) to a panel of either henipaviruses, influenza viruses, or sarbecoviruses
Neutralizing activity of plasma samples against known immunodominant zoonotic viral proteins | Day 0 and 2 optional visits at least 30 days apart between Day 180-720
  Measured by circulating antigen-specific B cells constituting approximately 0.001%-0.005% total PBMCs
Isolate viral antigen-specific B cells for phenotyping and immunoglobulin sequencing | Day 0 and 2 optional visits at least 30 days apart between Day 180-720
  Measured by isolation of an expected 20 million PBMCs from whole blood samples, yielding approximately 100-500 antigen-specific B cells for single-cell B-cell sequencing (anticipated cell death up to 50% during the isolation and sorting process)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Yek, MD, Principal Investigator — NIH/NIAID/Laboratory of Malaria and Vector Research (LMVR); Lon Chanthap, MD, Principal Investigator — Malaria Vector & Research Laboratory (MVRL) International Center of Excellence in Research Cambodia; Ly Sovann, MD, MTCM, Principal Investigator — Cambodian Center for Communicable Disease (CCDC) Ministry of Health, Cambodia
Locations (5):
- Cambodia (5):
  - Communicable Disease Control Department, Battambang
  - Communicable Disease Control Department, Kampong Thom
  - Communicable Disease Control Department, Kampot
  - Communicable Disease Control Department, Stung Treng
  - Communicable Disease Control Department, Takeo

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested from other researchers 5 years following completion of the primary endpoint by contacting the Principal Investigators.
Supporting Information: Study Protocol, CSR
Time Frame: 5 years following completion of the primary endpoint
Access Criteria: Researchers should contact the Principal Investigators with data requests.